CLINICAL TRIAL: NCT01277029
Title: Study of Psychiatric Aspects in Women With Lower Urinary Tract Symptoms
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 099022-E
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2021-06

CONDITIONS: Psychiatric Aspects in Women With Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- lower urinary tract symptoms
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — Psychopathology, personality traits of patients with lower urinary tract symptoms

SUMMARY:
To identify the differences in psychopathology, personality traits among different female LUTS subtypes.

ELIGIBILITY:
Inclusion Criteria:

* all cases with lower urinary tract symptoms

Exclusion Criteria:

* nil

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with low urinary tract symptoms
Sampling Method: Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan